CLINICAL TRIAL: NCT05469997
Title: Ketogenic Diet Interventions in Parkinson's Disease: Safeguarding the Gut Microbiome
Acronym: KIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Weston Family Foundation (Other)
Responsible Party: Principal Investigator, Silke Cresswell, Associate Professor (Tenure), University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H21-03747
Record Dates: First submitted 2022-06-15; First posted 2022-07-22 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Gut Microbiome; Ketogenic Diet; Mediterranean Diet; Medium-Chain Triglyceride; Life-style Interventions
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This safety study consists of two 8-week interventions (MeDi-MCT and MeDi-KD) in randomized order using a cross-over design, separated by an 8-week washout period. Participants will be randomized into either the MeDi-MCT or the MeDi-KD group for the first phase of the study. After 8-weeks of intervention, they will undergo an 8-week washout period where no interventions will be applied. Subsequently, the participants will commence the second phase of the study by receiving the other study intervention for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MeDi(KD-MCT) (Experimental): The participants in this arm will first undergo the MeDi-KD intervention followed by the MeDi-MCT intervention, after an 8-week washout period.
  Interventions: Behavioral: Mediterranean-Ketogenic Diet; Dietary Supplement: Mediterranean diet supplemented with medium-chain triglyceride oil
- MeDi(MCT-KD) (Experimental): The participants in this arm will first undergo the MeDi-MCT intervention followed by the MeDi-KD intervention, after an 8-week washout period.
  Interventions: Behavioral: Mediterranean-Ketogenic Diet; Dietary Supplement: Mediterranean diet supplemented with medium-chain triglyceride oil

INTERVENTIONS:
Behavioral: Mediterranean-Ketogenic Diet — In the MeDi-KD group, the participants will adhere to a modified Mediterranean-ketogenic diet. The ketogenic component of the diet will require limiting the intake of carbohydrates to about 10% of all calories consumed in a day, while obtaining most of the energy from healthy fats, mostly from plant-based sources (~70-75% of your daily caloric intake) and lean proteins (~15-20% of your daily caloric intake). The ketogenic ratio (the ratio of fat to carbohydrates) will be gradually increased during the first week from 1:1 to 3:1. The Mediterranean component of the diet will encourage the participants to consume more green leafy vegetables, nuts, and olive oil, while limiting the consumption of processed or fried food, red meat, full-fat dairy, and sweets.
  Other Names: MeDi-KD
Dietary Supplement: Mediterranean diet supplemented with medium-chain triglyceride oil — The participants will adhere to the Mediterranean diet. In addition, they will be asked to take two daily doses of medium-chain triglyceride oil (MCT oil).
  The MCT oil supplement (Nutiva MCT oil, Nutiva Inc.) is approved by Health Canada (NPN: 80086912) and will be used according to its approved condition of use (i.e., source of medium-chain fatty acids which supports energy production in the body at a cellular level [ATP]). Each serving of this product provides 130 Calories from MCTs (14 g) with a C8-C10 ratio of 60:40. Nutiva MCT oil can be mixed into any beverage of choice, but cannot be used for cooking.
  participants will start the intervention by taking 5 mL of MCT oil twice daily for the first day to acclimate their bodies to the supplement and gradually increase the dose to 14 g BID by the end of week 1. The participants may be asked to increase the dose to 20 mL of MCT twice daily if tolerability remains positive.
  Other Names: MeDi-MCT

SUMMARY:
Parkinson's Disease (PD) is the second most common neurodegenerative disorder with common gut-related symptoms, which are attributed to alterations in the gut microbiome - the collection of microorganisms that live within the gut. Classical ketogenic diets (KD) have shown to be beneficial in PD and non-PD populations but are associated with alterations in the gut microbiome that are characteristic of a perturbed system. This study aims to investigate the safety of modified Mediterranean-ketogenic interventions that are thought to be safer alternatives to the classical KD, as it relates to the gut microbiome health in patients with PD. We hypothesize that the modified Mediterranean-ketogenic interventions will not be associated with any significant perturbation of the gut microbiome in PD patients.

DETAILED DESCRIPTION:
Background:

Parkinson's disease (PD), the second most common and the most rapidly growing neurodegenerative disease worldwide [1,2]. Gut-related symptoms are common and often the initial symptoms, suggesting a possible intestinal origin of PD [4]. Over a dozen studies have demonstrated gut dysbiosis in PD with reduced diversity, increased pro-inflammatory capacity, and decreased Short-Chain Fatty Acids (SCFA) production as key characteristics [5-10] and persistently increased relative abundance of Akkermansia [5-17].

Emerging evidence suggests that both ketogenic [18-23] and Mediterranean diets [24-30] have beneficial and likely complementary effects in PD. Mediterranean diets (MeDi) are primarily but not exclusively plant-based [24]. Their promotion of high fiber content intake promotes the production of SCFA and are associated with improved gut microbiome health [25]. Ketogenic diets (KD) are high in fat, adequate in protein and very low in carbohydrates [31]. KD can provide ketone bodies (KB) [32] as an alternative fuel source to glucose, the utilization of which is perturbed in the PD brain [33]. Another method for inducing the state of ketosis is by consumption of ketogenic medium-chain triglycerides (MCTs) [43]. MCTs are converted to KBs, which can readily cross the blood-brain barrier and be used as an energy source [43]. Pilot trials in PD report improved Unified Parkinson's Disease Rating Scale (UPDRS) scores [20], cognitive performance [21] and non-motor symptoms [22] with KD interventions [23].

Several studies of classical KDs in non-PD populations have observed significant alterations in the gut microbiome, including an increase in Akkermansia [47] and a decrease in fecal SCFA levels [50].

By combining the principles of MeDi with ketogenic interventions, we hope to leverage the gut-health promoting aspects of the former with bioenergetics benefits of the latter, in a safe manner. To the best of our knowledge, no clinical trials have been performed into combined ketogenic and Medi-stye dietary interventions in PD yet.

Design:

A proof of concept, random order, cross-over study in participants with PD examining two 8-week interventions: (1) the Mediterranean ketogenic diet (MeDi-KD) and (2) the Mediterranean diet supplemented with medium-chain triglycerides (MeDi-MCT), separated by an 8-week washout period.

Hypothesis:

1. Neither the MeDi-MCT nor the MeDi-KD (pre-post comparison) will be significantly associated with measures of gut microbiome dysbiosis such as increased gut inflammation, impaired gut-barrier integrity, and reduced SCFA content.
2. Retention rates for both diets will be at least 75%.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-85 years
* PD diagnosis based on Movement Disorder Society (MDS) criteria [52]
* Hoehn & Yahr score of 1 to 3
* On stable dopaminergic medication for at least one month

Exclusion Criteria:

* Atypical parkinsonism
* Medical or psychiatric conditions that would prevent full participation in the nutrition intervention
* Significant dysphagia
* Diabetes on insulin
* Anti-coagulation on warfarin
* Inflammatory bowel disease
* Dementia defined by Montreal Cognitive Assessment (MoCA) Scores of less than 21
* Inability to fill in electronic questionnaires or understand study instructions
* Use of immunomodulatory agents
* Probiotic use in the last 4 weeks (except for dietary sources such as yoghurt, kefir etc.), or antibiotic use in the last 3 months prior to the trial
* Use of MCT oil or on ketogenic diet in last 8 weeks prior to the trial
* Allergic to MCT oil, coconut oil, or coconut

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline and difference across interventions in measures of fecal and serum calprotectin, a biomarker for gut inflammation. | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  We will assess changes from baseline in levels of fecal and serum calprotectin, a biomarker for gut inflammation that is found at elevated levels in PD patients, before and after each 8-week intervention. We will also compare the two interventions to determine their relative safety.
Changes from baseline and differences across interventions in other measures of gut health, namely short-chain fatty acid production, gut-barrier integrity, and microbial composition. | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  We will assess changes from baseline in the following biomarkers of gut health before and after each 8-week intervention:
  Short-chain fatty acid (SCFA)/ butyrate production measured in freshly frozen fecal samples Gut microbiome compositions measure in fecal samples. Levels of zonulin, a biomarker for gut-barrier function, measured in fecal and blood serum samples.
  We will track any potential adverse events.

SECONDARY OUTCOMES:
The number of participants who completed the study after successful enrollment relative to the total enrolled participants. | Post-intervention 1 (Week 8)/Post-intervention 2 (Week 24)
  We will assess the retention rate of participants with respect to each intervention to determine the feasibility of the proposed dietary interventions.
Percent time spent in clinically relevant levels of ketosis ( equivalent to >0.5 mmol/L) by each participant throughout each intervention. | Post-intervention 1 (Week 8)/Post-intervention 2 (Week 24)
  Adherence to the ketogenic dietary interventions will be measured using breath ketone analyzers (Ketonix). The participants will take daily measurements of their breath ketone levels and record them in their study journal.
  Percent time is determined by the number of days they successfully reach clinically relevant levels of ketosis relative to the total intervention days for each intervention (i.e. 56 days).

OTHER OUTCOMES:
Changes from baseline in motor and non-motor Parkinson's Disease symptoms after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Tracking changes from baseline in motor and non-motor Parkinson's disease symptoms using the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Tracking changes from baseline in severity of Fatigue Symptoms after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Tracking changes from baseline in severity of fatigue symptoms in the study participants using the Fatigue Severity Scale (FSS).
Changes from baseline in apathy symptoms after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Using Starkstein Apathy Scale (AS) to track changes from baseline in Apathy symptoms in the study participants after each intervention
Changes from baseline in depressive symptoms after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Using the Beck Depression Inventory II (BDI-II) to track changes in depressive symptoms from baseline in the study participants after each intervention
Changes from baseline in Anxiety symptoms after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Using the Parkinson's Anxiety Scale (PAS) to track changes in anxiety symptoms from baseline in the study participants after each intervention.
Tracking changes in the quality of life of the study participants after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Using the Parkinson's disease questionnaire (PDQ-39) to assess changes from baseline in the quality of life of the study participants after each intervention
Assessing changes in capacity for performing physical activities in the study participants after each intervention | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Physical Activity Scale for Individuals with Physical Disabilities (PASIPD)
Assessing changes in the the stool consistency of the study participants after each intervention | 24 weeks (weeks 1-24)
  Using Bristol Stool Chart to track the stool consistency of the study participants as they continue adhering to the study interventions.
Assessing the constipation and irritable bowl symptoms in the study participants | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Using the Rome III module to track changes from baseline in constipation and irritable bowel symptoms of the study participants after each intervention.
Determining the dietary habits of the study participants prior to beginning of the study | Preintervention 1 (Baseline 1)
  Using the Canadian version of the Diet History questionnaire (C-DHQ II) to determine the dietary habits of study participants prior to beginning of the study
Tracking changes in the cognitive function of the study participants | Preintervention 1 (Baseline 1)/ Post-intervention 1 (Week 8)/ Pre-intervention 2 (baseline 2; Week 16)/ Post-intervention 2 (Week 24)
  Using the National Health Institute Toolbox-Cognitive battery (NIHTB-CB) to assess changes from baseline in the cognitive function of the study participants after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Appel-Cresswell, MD, Principal Investigator — University of British Columbia
Locations (1):
- Djawad Mowafaghian Centre for Brain Health, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2016 Parkinson's Disease Collaborators. Global, regional, and national burden of Parkinson's disease, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):939-953. doi: 10.1016/S1474-4422(18)30295-3. Epub 2018 Oct 1. PMID 30287051
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] van der Kolk NM, de Vries NM, Kessels RPC, Joosten H, Zwinderman AH, Post B, Bloem BR. Effectiveness of home-based and remotely supervised aerobic exercise in Parkinson's disease: a double-blind, randomised controlled trial. Lancet Neurol. 2019 Nov;18(11):998-1008. doi: 10.1016/S1474-4422(19)30285-6. Epub 2019 Sep 11. PMID 31521532
- [Background] Borghammer P, Van Den Berge N. Brain-First versus Gut-First Parkinson's Disease: A Hypothesis. J Parkinsons Dis. 2019;9(s2):S281-S295. doi: 10.3233/JPD-191721. PMID 31498132
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Aho VTE, Houser MC, Pereira PAB, Chang J, Rudi K, Paulin L, Hertzberg V, Auvinen P, Tansey MG, Scheperjans F. Relationships of gut microbiota, short-chain fatty acids, inflammation, and the gut barrier in Parkinson's disease. Mol Neurodegener. 2021 Feb 8;16(1):6. doi: 10.1186/s13024-021-00427-6. PMID 33557896
- [Background] Hirayama M, Ohno K. Parkinson's Disease and Gut Microbiota. Ann Nutr Metab. 2021;77 Suppl 2:28-35. doi: 10.1159/000518147. Epub 2021 Sep 9. PMID 34500451
- [Background] Boertien JM, Pereira PAB, Aho VTE, Scheperjans F. Increasing Comparability and Utility of Gut Microbiome Studies in Parkinson's Disease: A Systematic Review. J Parkinsons Dis. 2019;9(s2):S297-S312. doi: 10.3233/JPD-191711. PMID 31498131
- [Background] Cirstea MS, Yu AC, Golz E, Sundvick K, Kliger D, Radisavljevic N, Foulger LH, Mackenzie M, Huan T, Finlay BB, Appel-Cresswell S. Microbiota Composition and Metabolism Are Associated With Gut Function in Parkinson's Disease. Mov Disord. 2020 Jul;35(7):1208-1217. doi: 10.1002/mds.28052. Epub 2020 May 1. PMID 32357258
- [Background] Wallen ZD, Appah M, Dean MN, Sesler CL, Factor SA, Molho E, Zabetian CP, Standaert DG, Payami H. Characterizing dysbiosis of gut microbiome in PD: evidence for overabundance of opportunistic pathogens. NPJ Parkinsons Dis. 2020 Jun 12;6:11. doi: 10.1038/s41531-020-0112-6. eCollection 2020. PMID 32566740
- [Background] Barichella M, Severgnini M, Cilia R, Cassani E, Bolliri C, Caronni S, Ferri V, Cancello R, Ceccarani C, Faierman S, Pinelli G, De Bellis G, Zecca L, Cereda E, Consolandi C, Pezzoli G. Unraveling gut microbiota in Parkinson's disease and atypical parkinsonism. Mov Disord. 2019 Mar;34(3):396-405. doi: 10.1002/mds.27581. Epub 2018 Dec 21. PMID 30576008
- [Background] Nishiwaki H, Ito M, Ishida T, Hamaguchi T, Maeda T, Kashihara K, Tsuboi Y, Ueyama J, Shimamura T, Mori H, Kurokawa K, Katsuno M, Hirayama M, Ohno K. Meta-Analysis of Gut Dysbiosis in Parkinson's Disease. Mov Disord. 2020 Sep;35(9):1626-1635. doi: 10.1002/mds.28119. Epub 2020 Jun 18. PMID 32557853
- [Background] Scheperjans F, Aho V, Pereira PA, Koskinen K, Paulin L, Pekkonen E, Haapaniemi E, Kaakkola S, Eerola-Rautio J, Pohja M, Kinnunen E, Murros K, Auvinen P. Gut microbiota are related to Parkinson's disease and clinical phenotype. Mov Disord. 2015 Mar;30(3):350-8. doi: 10.1002/mds.26069. Epub 2014 Dec 5. PMID 25476529
- [Background] Keshavarzian A, Green SJ, Engen PA, Voigt RM, Naqib A, Forsyth CB, Mutlu E, Shannon KM. Colonic bacterial composition in Parkinson's disease. Mov Disord. 2015 Sep;30(10):1351-60. doi: 10.1002/mds.26307. Epub 2015 Jul 16. PMID 26179554
- [Background] Unger MM, Spiegel J, Dillmann KU, Grundmann D, Philippeit H, Burmann J, Fassbender K, Schwiertz A, Schafer KH. Short chain fatty acids and gut microbiota differ between patients with Parkinson's disease and age-matched controls. Parkinsonism Relat Disord. 2016 Nov;32:66-72. doi: 10.1016/j.parkreldis.2016.08.019. Epub 2016 Aug 26. PMID 27591074
- [Background] Hill-Burns EM, Debelius JW, Morton JT, Wissemann WT, Lewis MR, Wallen ZD, Peddada SD, Factor SA, Molho E, Zabetian CP, Knight R, Payami H. Parkinson's disease and Parkinson's disease medications have distinct signatures of the gut microbiome. Mov Disord. 2017 May;32(5):739-749. doi: 10.1002/mds.26942. Epub 2017 Feb 14. PMID 28195358
- [Background] Heintz-Buschart A, Pandey U, Wicke T, Sixel-Doring F, Janzen A, Sittig-Wiegand E, Trenkwalder C, Oertel WH, Mollenhauer B, Wilmes P. The nasal and gut microbiome in Parkinson's disease and idiopathic rapid eye movement sleep behavior disorder. Mov Disord. 2018 Jan;33(1):88-98. doi: 10.1002/mds.27105. Epub 2017 Aug 26. PMID 28843021
- [Background] Wlodarek D. Role of Ketogenic Diets in Neurodegenerative Diseases (Alzheimer's Disease and Parkinson's Disease). Nutrients. 2019 Jan 15;11(1):169. doi: 10.3390/nu11010169. PMID 30650523
- [Background] Paoli A, Bianco A, Damiani E, Bosco G. Ketogenic diet in neuromuscular and neurodegenerative diseases. Biomed Res Int. 2014;2014:474296. doi: 10.1155/2014/474296. Epub 2014 Jul 3. PMID 25101284
- [Background] Vanitallie TB, Nonas C, Di Rocco A, Boyar K, Hyams K, Heymsfield SB. Treatment of Parkinson disease with diet-induced hyperketonemia: a feasibility study. Neurology. 2005 Feb 22;64(4):728-30. doi: 10.1212/01.WNL.0000152046.11390.45. PMID 15728303
- [Background] Krikorian R, Shidler MD, Summer SS, Sullivan PG, Duker AP, Isaacson RS, Espay AJ. Nutritional ketosis for mild cognitive impairment in Parkinson's disease: A controlled pilot trial. Clin Park Relat Disord. 2019 Aug 6;1:41-47. doi: 10.1016/j.prdoa.2019.07.006. eCollection 2019. PMID 34316598
- [Background] Phillips MCL, Murtagh DKJ, Gilbertson LJ, Asztely FJS, Lynch CDP. Low-fat versus ketogenic diet in Parkinson's disease: A pilot randomized controlled trial. Mov Disord. 2018 Aug;33(8):1306-1314. doi: 10.1002/mds.27390. Epub 2018 Aug 11. PMID 30098269
- [Background] Choi A, Hallett M, Ehrlich D. Nutritional Ketosis in Parkinson's Disease - a Review of Remaining Questions and Insights. Neurotherapeutics. 2021 Jul;18(3):1637-1649. doi: 10.1007/s13311-021-01067-w. Epub 2021 Jul 7. PMID 34235637
- [Background] Davis C, Bryan J, Hodgson J, Murphy K. Definition of the Mediterranean Diet; a Literature Review. Nutrients. 2015 Nov 5;7(11):9139-53. doi: 10.3390/nu7115459. PMID 26556369
- [Background] Nagpal R, Shively CA, Register TC, Craft S, Yadav H. Gut microbiome-Mediterranean diet interactions in improving host health. F1000Res. 2019 May 21;8:699. doi: 10.12688/f1000research.18992.1. eCollection 2019. PMID 32704349
- [Background] Alcalay RN, Gu Y, Mejia-Santana H, Cote L, Marder KS, Scarmeas N. The association between Mediterranean diet adherence and Parkinson's disease. Mov Disord. 2012 May;27(6):771-4. doi: 10.1002/mds.24918. Epub 2012 Feb 7. PMID 22314772
- [Background] Maraki MI, Yannakoulia M, Stamelou M, Stefanis L, Xiromerisiou G, Kosmidis MH, Dardiotis E, Hadjigeorgiou GM, Sakka P, Anastasiou CA, Simopoulou E, Scarmeas N. Mediterranean diet adherence is related to reduced probability of prodromal Parkinson's disease. Mov Disord. 2019 Jan;34(1):48-57. doi: 10.1002/mds.27489. Epub 2018 Oct 10. PMID 30306634
- [Background] Agarwal P, Wang Y, Buchman AS, Holland TM, Bennett DA, Morris MC. MIND Diet Associated with Reduced Incidence and Delayed Progression of ParkinsonismA in Old Age. J Nutr Health Aging. 2018;22(10):1211-1215. doi: 10.1007/s12603-018-1094-5. PMID 30498828
- [Background] Molsberry S, Bjornevik K, Hughes KC, Healy B, Schwarzschild M, Ascherio A. Diet pattern and prodromal features of Parkinson disease. Neurology. 2020 Oct 13;95(15):e2095-e2108. doi: 10.1212/WNL.0000000000010523. Epub 2020 Aug 19. PMID 32817391
- [Background] Metcalfe-Roach A, Yu AC, Golz E, Cirstea M, Sundvick K, Kliger D, Foulger LH, Mackenzie M, Finlay BB, Appel-Cresswell S. MIND and Mediterranean Diets Associated with Later Onset of Parkinson's Disease. Mov Disord. 2021 Apr;36(4):977-984. doi: 10.1002/mds.28464. Epub 2021 Jan 6. PMID 33404118
- [Background] Freeman JM, Kossoff EH, Hartman AL. The ketogenic diet: one decade later. Pediatrics. 2007 Mar;119(3):535-43. doi: 10.1542/peds.2006-2447. PMID 17332207
- [Background] Nylen K, Likhodii S, Burnham WM. The ketogenic diet: proposed mechanisms of action. Neurotherapeutics. 2009 Apr;6(2):402-5. doi: 10.1016/j.nurt.2009.01.021. PMID 19332336
- [Background] Norwitz NG, Hu MT, Clarke K. The Mechanisms by Which the Ketone Body D-beta-Hydroxybutyrate May Improve the Multiple Cellular Pathologies of Parkinson's Disease. Front Nutr. 2019 May 14;6:63. doi: 10.3389/fnut.2019.00063. eCollection 2019. PMID 31139630
- [Background] Cahill GF Jr. Fuel metabolism in starvation. Annu Rev Nutr. 2006;26:1-22. doi: 10.1146/annurev.nutr.26.061505.111258. PMID 16848698
- [Background] Owen OE, Morgan AP, Kemp HG, Sullivan JM, Herrera MG, Cahill GF Jr. Brain metabolism during fasting. J Clin Invest. 1967 Oct;46(10):1589-95. doi: 10.1172/JCI105650. PMID 6061736
- [Background] Shimazu T, Hirschey MD, Newman J, He W, Shirakawa K, Le Moan N, Grueter CA, Lim H, Saunders LR, Stevens RD, Newgard CB, Farese RV Jr, de Cabo R, Ulrich S, Akassoglou K, Verdin E. Suppression of oxidative stress by beta-hydroxybutyrate, an endogenous histone deacetylase inhibitor. Science. 2013 Jan 11;339(6116):211-4. doi: 10.1126/science.1227166. Epub 2012 Dec 6. PMID 23223453
- [Background] Gasior M, Rogawski MA, Hartman AL. Neuroprotective and disease-modifying effects of the ketogenic diet. Behav Pharmacol. 2006 Sep;17(5-6):431-9. doi: 10.1097/00008877-200609000-00009. PMID 16940764
- [Background] Garcia-Rodriguez D, Gimenez-Cassina A. Ketone Bodies in the Brain Beyond Fuel Metabolism: From Excitability to Gene Expression and Cell Signaling. Front Mol Neurosci. 2021 Aug 27;14:732120. doi: 10.3389/fnmol.2021.732120. eCollection 2021. PMID 34512261
- [Background] D'Andrea Meira I, Romao TT, Pires do Prado HJ, Kruger LT, Pires MEP, da Conceicao PO. Ketogenic Diet and Epilepsy: What We Know So Far. Front Neurosci. 2019 Jan 29;13:5. doi: 10.3389/fnins.2019.00005. eCollection 2019. PMID 30760973
- [Background] Yuan X, Wang J, Yang S, Gao M, Cao L, Li X, Hong D, Tian S, Sun C. Effect of the ketogenic diet on glycemic control, insulin resistance, and lipid metabolism in patients with T2DM: a systematic review and meta-analysis. Nutr Diabetes. 2020 Nov 30;10(1):38. doi: 10.1038/s41387-020-00142-z. PMID 33257645
- [Background] Castellana M, Conte E, Cignarelli A, Perrini S, Giustina A, Giovanella L, Giorgino F, Trimboli P. Efficacy and safety of very low calorie ketogenic diet (VLCKD) in patients with overweight and obesity: A systematic review and meta-analysis. Rev Endocr Metab Disord. 2020 Mar;21(1):5-16. doi: 10.1007/s11154-019-09514-y. PMID 31705259
- [Background] Myette-Cote E, Soto-Mota A, Cunnane SC. Ketones: potential to achieve brain energy rescue and sustain cognitive health during ageing. Br J Nutr. 2022 Aug 14;128(3):407-423. doi: 10.1017/S0007114521003883. Epub 2021 Sep 28. PMID 34581265
- [Background] Marten B, Pfeuffer M, Schrezenmeir J. Medium-chain triglycerides. International Dairy Journal. 2006;16(11):1374-1382. doi:10.1016/j.idairyj.2006.06.015
- [Background] Neal EG, Chaffe H, Schwartz RH, Lawson MS, Edwards N, Fitzsimmons G, Whitney A, Cross JH. A randomized trial of classical and medium-chain triglyceride ketogenic diets in the treatment of childhood epilepsy. Epilepsia. 2009 May;50(5):1109-17. doi: 10.1111/j.1528-1167.2008.01870.x. Epub 2008 Nov 19. PMID 19054400
- [Background] Fortier M, Castellano CA, St-Pierre V, Myette-Cote E, Langlois F, Roy M, Morin MC, Bocti C, Fulop T, Godin JP, Delannoy C, Cuenoud B, Cunnane SC. A ketogenic drink improves cognition in mild cognitive impairment: Results of a 6-month RCT. Alzheimers Dement. 2021 Mar;17(3):543-552. doi: 10.1002/alz.12206. Epub 2020 Oct 26. PMID 33103819
- [Background] Fortier M, Castellano CA, Croteau E, Langlois F, Bocti C, St-Pierre V, Vandenberghe C, Bernier M, Roy M, Descoteaux M, Whittingstall K, Lepage M, Turcotte EE, Fulop T, Cunnane SC. A ketogenic drink improves brain energy and some measures of cognition in mild cognitive impairment. Alzheimers Dement. 2019 May;15(5):625-634. doi: 10.1016/j.jalz.2018.12.017. Epub 2019 Apr 23. PMID 31027873
- [Background] Paoli A, Mancin L, Bianco A, Thomas E, Mota JF, Piccini F. Ketogenic Diet and Microbiota: Friends or Enemies? Genes (Basel). 2019 Jul 15;10(7):534. doi: 10.3390/genes10070534. PMID 31311141
- [Background] Nagpal R, Neth BJ, Wang S, Craft S, Yadav H. Modified Mediterranean-ketogenic diet modulates gut microbiome and short-chain fatty acids in association with Alzheimer's disease markers in subjects with mild cognitive impairment. EBioMedicine. 2019 Sep;47:529-542. doi: 10.1016/j.ebiom.2019.08.032. Epub 2019 Aug 30. PMID 31477562
- [Background] Olson CA, Vuong HE, Yano JM, Liang QY, Nusbaum DJ, Hsiao EY. The Gut Microbiota Mediates the Anti-Seizure Effects of the Ketogenic Diet. Cell. 2018 Jun 14;173(7):1728-1741.e13. doi: 10.1016/j.cell.2018.04.027. Epub 2018 May 24. PMID 29804833
- [Background] Ferraris C, Meroni E, Casiraghi MC, Tagliabue A, De Giorgis V, Erba D. One Month of Classic Therapeutic Ketogenic Diet Decreases Short Chain Fatty Acids Production in Epileptic Patients. Front Nutr. 2021 Mar 29;8:613100. doi: 10.3389/fnut.2021.613100. eCollection 2021. PMID 33855040
- [Background] Ang QY, Alexander M, Newman JC, Tian Y, Cai J, Upadhyay V, Turnbaugh JA, Verdin E, Hall KD, Leibel RL, Ravussin E, Rosenbaum M, Patterson AD, Turnbaugh PJ. Ketogenic Diets Alter the Gut Microbiome Resulting in Decreased Intestinal Th17 Cells. Cell. 2020 Jun 11;181(6):1263-1275.e16. doi: 10.1016/j.cell.2020.04.027. Epub 2020 May 20. PMID 32437658
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] van Delft R, Lambrechts D, Verschuure P, Hulsman J, Majoie M. Blood beta-hydroxybutyrate correlates better with seizure reduction due to ketogenic diet than do ketones in the urine. Seizure. 2010 Jan;19(1):36-9. doi: 10.1016/j.seizure.2009.10.009. Epub 2009 Dec 3. PMID 19962324
- [Background] Anderson JC, Mattar SG, Greenway FL, Lindquist RJ. Measuring ketone bodies for the monitoring of pathologic and therapeutic ketosis. Obes Sci Pract. 2021 May 4;7(5):646-656. doi: 10.1002/osp4.516. eCollection 2021 Oct. PMID 34631141
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Wood DE, Lu J, Langmead B. Improved metagenomic analysis with Kraken 2. Genome Biol. 2019 Nov 28;20(1):257. doi: 10.1186/s13059-019-1891-0. PMID 31779668
- [Background] Silva GG, Green KT, Dutilh BE, Edwards RA. SUPER-FOCUS: a tool for agile functional analysis of shotgun metagenomic data. Bioinformatics. 2016 Feb 1;32(3):354-61. doi: 10.1093/bioinformatics/btv584. Epub 2015 Oct 9. PMID 26454280
- [Background] Zheng X, Qiu Y, Zhong W, Baxter S, Su M, Li Q, Xie G, Ore BM, Qiao S, Spencer MD, Zeisel SH, Zhou Z, Zhao A, Jia W. A targeted metabolomic protocol for short-chain fatty acids and branched-chain amino acids. Metabolomics. 2013 Aug 1;9(4):818-827. doi: 10.1007/s11306-013-0500-6. PMID 23997757
- [Background] Schwiertz A, Spiegel J, Dillmann U, Grundmann D, Burmann J, Fassbender K, Schafer KH, Unger MM. Fecal markers of intestinal inflammation and intestinal permeability are elevated in Parkinson's disease. Parkinsonism Relat Disord. 2018 May;50:104-107. doi: 10.1016/j.parkreldis.2018.02.022. Epub 2018 Feb 12. PMID 29454662
- [Background] Dumitrescu L, Marta D, Danau A, Lefter A, Tulba D, Cozma L, Manole E, Gherghiceanu M, Ceafalan LC, Popescu BO. Serum and Fecal Markers of Intestinal Inflammation and Intestinal Barrier Permeability Are Elevated in Parkinson's Disease. Front Neurosci. 2021 Jun 18;15:689723. doi: 10.3389/fnins.2021.689723. eCollection 2021. PMID 34220443
- [Background] Ohlsson B, Roth B, Larsson E, Hoglund P. Calprotectin in serum and zonulin in serum and feces are elevated after introduction of a diet with lower carbohydrate content and higher fiber, fat and protein contents. Biomed Rep. 2017 Apr;6(4):411-422. doi: 10.3892/br.2017.865. Epub 2017 Feb 22. PMID 28413639
- [Background] Harms AS, Ferreira SA, Romero-Ramos M. Periphery and brain, innate and adaptive immunity in Parkinson's disease. Acta Neuropathol. 2021 Apr;141(4):527-545. doi: 10.1007/s00401-021-02268-5. Epub 2021 Feb 8. PMID 33555429
- [Background] Tran HQ, Bretin A, Adeshirlarijaney A, Yeoh BS, Vijay-Kumar M, Zou J, Denning TL, Chassaing B, Gewirtz AT. "Western Diet"-Induced Adipose Inflammation Requires a Complex Gut Microbiota. Cell Mol Gastroenterol Hepatol. 2020;9(2):313-333. doi: 10.1016/j.jcmgh.2019.09.009. Epub 2019 Oct 5. PMID 31593782
- [Background] Chrysohoou C, Panagiotakos DB, Pitsavos C, Das UN, Stefanadis C. Adherence to the Mediterranean diet attenuates inflammation and coagulation process in healthy adults: The ATTICA Study. J Am Coll Cardiol. 2004 Jul 7;44(1):152-8. doi: 10.1016/j.jacc.2004.03.039. PMID 15234425
- [Background] Sawada H, Oeda T, Umemura A, Tomita S, Kohsaka M, Park K, Yamamoto K, Sugiyama H. Baseline C-Reactive Protein Levels and Life Prognosis in Parkinson Disease. PLoS One. 2015 Jul 28;10(7):e0134118. doi: 10.1371/journal.pone.0134118. eCollection 2015. PMID 26218286
- [Background] Umemura A, Oeda T, Yamamoto K, Tomita S, Kohsaka M, Park K, Sugiyama H, Sawada H. Baseline Plasma C-Reactive Protein Concentrations and Motor Prognosis in Parkinson Disease. PLoS One. 2015 Aug 26;10(8):e0136722. doi: 10.1371/journal.pone.0136722. eCollection 2015. PMID 26308525
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Brown RG, Dittner A, Findley L, Wessely SC. The Parkinson fatigue scale. Parkinsonism Relat Disord. 2005 Jan;11(1):49-55. doi: 10.1016/j.parkreldis.2004.07.007. PMID 15619463
- [Background] Starkstein SE, Mayberg HS, Preziosi TJ, Andrezejewski P, Leiguarda R, Robinson RG. Reliability, validity, and clinical correlates of apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 1992 Spring;4(2):134-9. doi: 10.1176/jnp.4.2.134. PMID 1627973
- [Background] Beck AT, Steer RA, Brown G. Beck Depression Inventory-II. Psychol Assess [Internet]. [doi: 10.1037/t00742-000]
- [Background] Leentjens AF, Dujardin K, Pontone GM, Starkstein SE, Weintraub D, Martinez-Martin P. The Parkinson Anxiety Scale (PAS): development and validation of a new anxiety scale. Mov Disord. 2014 Jul;29(8):1035-43. doi: 10.1002/mds.25919. Epub 2014 May 23. PMID 24862344
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Washburn RA, Zhu W, McAuley E, Frogley M, Figoni SF. The physical activity scale for individuals with physical disabilities: development and evaluation. Arch Phys Med Rehabil. 2002 Feb;83(2):193-200. doi: 10.1053/apmr.2002.27467. PMID 11833022
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Drossman DA, Dumitrascu DL. Rome III: New standard for functional gastrointestinal disorders. J Gastrointestin Liver Dis. 2006 Sep;15(3):237-41. PMID 17013448
- [Background] Thompson FE, Subar AF, Brown CC, Smith AF, Sharbaugh CO, Jobe JB, Mittl B, Gibson JT, Ziegler RG. Cognitive research enhances accuracy of food frequency questionnaire reports: results of an experimental validation study. J Am Diet Assoc. 2002 Feb;102(2):212-25. doi: 10.1016/s0002-8223(02)90050-7. PMID 11846115
- [Background] Heaton RK, Akshoomoff N, Tulsky D, Mungas D, Weintraub S, Dikmen S, Beaumont J, Casaletto KB, Conway K, Slotkin J, Gershon R. Reliability and validity of composite scores from the NIH Toolbox Cognition Battery in adults. J Int Neuropsychol Soc. 2014 Jul;20(6):588-98. doi: 10.1017/S1355617714000241. Epub 2014 Jun 24. PMID 24960398
- [Background] Nygaard HB, Kent BA, Stager S, et al. A phase 1B multiple ascending dose study of the safety, tolerability, pharmacokinetics, and pharmacodynamics of a medium chain triglyceride supplement in Alzheimer's disease: Brain energy rescue interventions to treat or delay Alzheimer's disease. Alzheimer's & Dementia. 2020;16(S10). doi:10.1002/alz.037960
- [Background] Ma D, Wang AC, Parikh I, Green SJ, Hoffman JD, Chlipala G, Murphy MP, Sokola BS, Bauer B, Hartz AMS, Lin AL. Ketogenic diet enhances neurovascular function with altered gut microbiome in young healthy mice. Sci Rep. 2018 Apr 27;8(1):6670. doi: 10.1038/s41598-018-25190-5. PMID 29703936
- [Background] Mufti A, Mirali S, Abduelmula A, McDonald KA, Alabdulrazzaq S, Sachdeva M, Yeung J. Clinical manifestations and treatment outcomes in prurigo pigmentosa (Nagashima disease): A systematic review of the literature. JAAD Int. 2021 Apr 10;3:79-87. doi: 10.1016/j.jdin.2021.03.003. eCollection 2021 Jun. PMID 34409375
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Derived] Tosefsky K, Lam JS, Wang YN, Keymanesh S, Kuan AJ, Metcalfe-Roach A, Cirstea MS, Sacheli MA, Brett Finlay B, Cohen TR, Appel-Cresswell S. A randomized safety and feasibility crossover trial of two Mediterranean-ketogenic interventions in individuals with Parkinson's disease. J Parkinsons Dis. 2026 Feb 4:1877718X261418986. doi: 10.1177/1877718X261418986. Online ahead of print. PMID 41637153
- [Derived] Tosefsky KN, Wang YN, Lam JS, Cohen TR, Appel-Cresswell S. Exploring the Facilitators and Barriers of Adherence to Mediterranean-Ketogenic Dietary Interventions in Parkinson's Disease: A Qualitative Study. Curr Dev Nutr. 2025 Oct 30;9(11):107591. doi: 10.1016/j.cdnut.2025.107591. eCollection 2025 Nov. PMID 41341605